CLINICAL TRIAL: NCT03036033
Title: The SaeboGlove Evaluation Trial in Stroke
Brief Title: The SaeboGlove Evaluation Trial
Acronym: T-SET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Jesse Dawson, Clinical Reader, NHS Greater Glasgow and Clyde
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: GN16ST162; Res16/A169 (Other Grant/Funding Number: CHSS); 16/NS/0112 (Other: North of Scotland Research Ethics Service); 207595 (Other: Integrated Research Application System)
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Stroke; Cerebral Vascular Disorder; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Single group, open feasibility study of use of a CE marked and available device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SaeboGlove Therapy (Experimental): All participants will be given a SaeboGlove for a 4-week period to use along side their routine functional based training program.
  Interventions: Device: SaeboGlove

INTERVENTIONS:
Device: SaeboGlove — All participants are given a Saebo glove to use during their stroke recovery.

SUMMARY:
This study evaluates the safety, feasibility and usability of a SaeboGlove rehabilitation device in the treatment of patients who have reduced ability to open their hand due to weakness after an acute stroke.

DETAILED DESCRIPTION:
The SaeboGlove is a new rehabilitation aid that can be used in people with hand weakness after a neurological injury. It assists the hand to open, which is crucial for people to grasp, and release everyday objects. It may improve function by doing this but may also help people with severe weakness take part more fully in therapy sessions. This glove is already marketed and is being used in some NHS sites. This trial will assess how it could be used in NHS practice in acute stroke patients and will develop a plan to implement this.

ELIGIBILITY:
Inclusion Criteria:

1. Able to consent
2. Aged ≥18 years
3. Diagnosis of stroke occurring ≤30 days ago
4. Reduced active range of movement wrist and / or finger extension
5. Modified ashworth score at wrist and fingers ≤ 2
6. Some initiation of gross active finger flexion
7. At least 10 degrees passive range of motion wrist extension
8. Considered able to learn to don / doff a SaeboGlove +/- help of willing carer
9. Ability to engage in some independent rehabilitation +/- help of willing carer
10. Considered able to comply with the requirements of protocol?

Exclusion Criteria:

1. Presence of >5-10 degrees digital contractures
2. Presence of other upper limb impairment that would influence participation (e.g. fixed contracture, frozen shoulder, severe arthritis or upper limb pain)
3. Presence of other conditions likely to influence participation (e.g. medically unstable, registered blind, terminal cancer, severe mood, cognitive or language issues)
4. Participating in another stroke rehabilitation trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-01-26 (Actual); Primary Completion 2017-05-25 (Estimated); Study Completion 2017-07-25 (Estimated)

PRIMARY OUTCOMES:
Number of sessions performed using the SaeboGlove | One month
  Feasibility

SECONDARY OUTCOMES:
Therapy Intensity | Cumulative over one month
  Number of movement repetitions performed using the SaeboGlove
Participant, Carer and Therapist Usability and Training Questionnaire | One month
  Bespoke questionnaire
Box and Block Test | One month
  Measure to assess gross dexterity
Action Research Arm Test (ARAT) | One month
  Measure to assess arm function
Motor Activity Log (MAL) | One month
  Interview intended to examine how much and how well the participant uses arm
Number of adverse events related to using the SaeboGlove | One month
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jesse Dawson, Principal Investigator — University of Glasgow
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No